CLINICAL TRIAL: NCT04545970
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Efficacy and Safety of an Anti-Aging Serum in the Treatment of Facial Lines
Brief Title: A Clinical Study to Evaluate Efficacy and Safety of a Cosmetic Product in the Treatment of Facial Lines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Collaborators: Ablon Skin Institute Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASIRC-RS-01
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Fine Lines; Wrinkles; Photoaging
Keywords: anti-aging; serum
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Investigator
Masking Description: Randomization will occur by assignment to either the active group or placebo group using a randomization table prepared prior to the start of the study by a non-participating staff member at the office of the investigator. Subjects will be assigned a number in numerical order as enrolled. The unblinded staff member will take a set of products from one of two groups of labeled active product vs. placebo and fill in the patient number and distribution date on the bottles to be dispensed to the subject.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-aging Serum (Active Comparator): Dosage form: Serum composed of water, thickener, and bioactive ingredients including antioxidants and peptides.
  Frequency of Dosage: Two times daily. Subjects are asked to pump 2x and apply on global face morning and evening.
  Study Duration: 12 weeks.
  Interventions: Combination Product: Facial cleanser; Combination Product: Facial moisturizer; Combination Product: Sunscreen
- Placebo Serum (Placebo Comparator): Dosage form: Serum composed of water and thickener. Frequency of Dosage: Two times daily. Subjects are asked to pump 2x and apply on global face morning and evening.
  Study Duration: 12 weeks.
  Interventions: Combination Product: Facial cleanser; Combination Product: Facial moisturizer; Combination Product: Sunscreen

INTERVENTIONS:
Combination Product: Facial cleanser — Facial cleanser to be used by study participants
Combination Product: Facial moisturizer — Bland moisturizer to be used by study participants after serum in the evening.
Combination Product: Sunscreen — Sunscreen to be applied after application of serum in the morning.
  Other Names: Neutrogena Sheer Zinc SPF 30

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial was conducted to assess the efficacy and safety of an anti-aging serum to improve the appearance of expression lines as well as overall skin health of aging skin after 12 weeks of twice-daily use in female subjects, aged 35-60, compared to placebo. A total of 55 subjects completed study participation which included 33 subjects in the active group and 22 subjects in the placebo group.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled clinical trial is being conducted to assess the efficacy and safety of the anti-aging serum when used over the course of 12 weeks by women with mild to moderate fine lines, wrinkles and overall photodamage on the global face.

Efficacy and tolerability will be assess through clinical grading at baseline, weeks 4, 8, and 12. Efficacy evaluation on fine lines and wrinkles through clinical grading will also be performed at 15 minutes post product application. Self-assessment questionnaires and VISIA photography will be completed at baseline, weeks 4, 8, and 12. 3D PRIMOS photography will be performed at baseline, weeks 8 and 12.

A total of 55 subjects completed study participation which included 33 subjects in the active group and 22 subjects in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 35 and 60 years were scheduled for eligibility screening at the study site.
* Women with Fitzpatrick Skin Type I-VI
* Subjects must have mild to moderate global face wrinkles and fine lines
* Subjects may have mild to moderate photo-aging secondary to physiologic aging
* Subjects must have no known medical conditions that, in the investigator's opinion, may interfere with study participation.
* Subjects must be willing to provide verbal understanding and written informed consent.

Exclusion Criteria:

* Female subjects who are pregnant, breast feeding, or planning a pregnancy.
* Subjects with severe overall photo damage as determined by the Investigator.
* Subjects who have any dermatological disorder, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's skin, including rosacea, acne, and excessively oily or dry skin.
* Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study products.
* Subjects use of any medications that are known to potentially cause changes in the facial skin as determined by the Investigator.
* Subjects who spend excessive time out in the sun.
* Subjects who are unwilling or unable to comply with the requirements of the protocol.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Clinical Efficacy Graded by Griffiths' Scale | 12 weeks
  The primary efficacy endpoint will be the Investigator Clinical Grading using Modified Griffith's 10-point Scale. A decrease in scores at Day 28, Day 56 and Day 84 in comparison to baseline indicates an improvement for the indicated parameter.The efficacy parameters will be assessed globally on each subject's face using a modified Griffiths' 10-point scale according to the following numerical definitions (half-point scores may be used as necessary to more accurately describe the skin condition):
  0 = none (best possible condition); 1 to 3 = mild; 4 to 6 = moderate;7 to 9 = severe (worst possible condition). The lower the score equates to the best possible outcome.
Objective Tolerability: scores | 12 weeks
  The primary tolerability endpoint will be the Investigator Tolerability Assessment of Erythema, Edema and Dryness. A decrease in scores or lack of significant increase at Day 28, Day 56 and Day 84 in comparison to Baseline indicates tolerability/safety of the test material. Four point scale with a lower score indicating a better outcome.
  Example for Erythema:Erythema 0 = None No erythema of the treatment area
  1. = Mild Slight, but definite redness of the treatment area
  2. = Moderate Definite redness of the treatment area
  3. = Severe Marked redness of the treatment area

SECONDARY OUTCOMES:
Subjective Tolerability: scores | 12 weeks
  The secondary tolerability endpoint will be the Subject Tolerability Assessment of Burning, Itching and Stinging. A decrease in scores or lack of significant increase at Day 28, Day 56 and Day 84 in comparison to Baseline indicates tolerability/safety of the test material. Four point scale with a lower score indicating a better outcome.
  Example Burning. 0 = None No burning of the treatment area
  1. = Mild Slight burning sensation of the treatment area; not really bothersome
  2. = Moderate Definite warm, burning of the treatment area that is somewhat bothersome.
  3. = Severe Hot burning sensation of the treatment area that causes definite discomfort and may interrupt daily activities and/or sleep
Self Assessment Questions | 12 weeks
  The secondary efficacy endpoints will be the Self-Assessment Questionnaire and the Subject Treatment Satisfaction and Ease of Use Questionnaire. A decrease or increase in response values at Day 28, Day 56 and Day 84 indicates an improvement compared to baseline response values. Subjects are asked to rate based on a scoring system of the following: from 5 (completely agree) to 1 (completely disagree). The best outcome is to Completely Agree with the statement/ question being asked.

CONTACTS AND LOCATIONS:
Overall Officials: Glynis Ablon, MD, FAAD, Principal Investigator — Ablon Skin Institute Research Center
Locations (1):
- Ablon Skin Institute Research Center, Manhattan Beach, California, United States